CLINICAL TRIAL: NCT04606797
Title: Targeting Mailed Nicotine Patch Distribution Interventions to Rural Regions of Canada: Randomized Controlled Trial
Brief Title: Targeting Mailed Nicotine Patch Distribution Interventions to Rural Regions of Canada
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 006/2020
Record Dates: First submitted 2020-10-24; First posted 2020-10-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotine Replacement Therapy (Experimental)
  Interventions: Drug: Nicotine patch
- Control (No Intervention)

INTERVENTIONS:
Drug: Nicotine patch — Nicotine transdermal patches as per product monograph
  Other Names: Nicoderm
  Arms: Nicotine Replacement Therapy

SUMMARY:
This study will examine the impact of mailed distribution of free Nicotine Replacement Therapy to smokers in rural regions. Telephone numbers will be randomly selected from across Canada in order to recruit adult smokers interested in completing a smoking survey and willing to be interviewed again in 6 months time. Study participants will be asked about their smoking history and a hypothetical question: would they be interested in receiving the nicotine patches if this were to be provided to them free of charge? Participants expressing interest will be randomly assigned to one of two groups. One group will be offered the opportunity to actually receive a program of 5 weeks of the nicotine patch for free right away and the other group will not be offered the free nicotine patches. The proportions of smokers in the two groups who quit smoking by the 6-month interview will be compared. Characteristics of the participants and the municipalities in which they live will be used to explain why the nicotine patch intervention has a larger impact in some rural regions compared to others

This projects seeks to determine the impact of mailed NRT intervention on increasing quit rates in rural areas. In addition, it seeks to understand the social determinants of health driving the large effects expected based on previous findings.

DETAILED DESCRIPTION:
Quitting smoking is the most effective way of reducing the risk of cancer. One way of helping people stop smoking is to provide them with free Nicotine Replacement Therapy (NRT; e.g., nicotine patch), such as when NRT is sent to people by postal mail as part of a mass distribution initiative. Our previous research indicated that the impact of the mailed NRT intervention on increasing quit rates in rural areas may be substantial. The current research project seeks to confirm this finding and to understand the social determinants of health driving these anticipated large effects. This information is essential in order to target limited health resources to regions that are most in need, and who are likely to experience the greatest benefit.

A two-stage recruitment process will be employed, in the context of a general population survey with a 6-month follow-up. Random digit dialling of telephone numbers from rural regions of Canada will identify households with adult (age 18 or over) smokers who smoke 10 or more cigarettes a day and who are willing to take part in a smoking study that involves two interviews. Residence of participants in rural regions will be confirmed by postal code matching. As part of the baseline survey, eligible subjects will be identified for the second recruitment - randomization of smokers into experimental and control conditions to be offered versus not offered Nicotine Patches. A randomized half of the eligible participants will be assigned to the experimental condition and asked for their permission to have Nicotine Patches sent to their home. The 6-month follow-up survey will be conducted 6-months after the baseline survey.

The primary hypothesis is that participants receiving the NRT package will display significantly greater quit rates (30 day abstinence) at 6-month follow-up as compared to those not offered the NRT package.

ELIGIBILITY:
Inclusion Criteria:

* Smoke 10 or more cigarettes per day
* Willing to be interviewed at baseline and 6 months
* Interest in using nicotine patch to quit smoking
* Intent to use nicotine patch within 1 week of receipt
* Willing to have nicotine patches sent to their home

Exclusion Criteria:

* Contraindication to NRT patch use (e.g. pregnant, intending on becoming pregnant, allergic to tape, serious heart circulation problem, not including high blood pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
30-day point prevalence abstinence | 6 month follow-up
  Self-reported no smoking of cigarettes in the past 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Cunningham John, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Cunningham JA, Chaiton M, Leatherdale ST, Godinho A, Schell C. Effect of Postal-Mailed Nicotine Patches on Tobacco Cessation Among Smokers in Rural Canada: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2325206. doi: 10.1001/jamanetworkopen.2023.25206. PMID 37486633
- [Derived] Cunningham JA, Chaiton M, Leatherdale ST, Godinho A, Schell C. Targeting mailed nicotine patch distribution interventions to rural regions of Canada: protocol for a randomized controlled trial. BMC Public Health. 2020 Nov 23;20(1):1757. doi: 10.1186/s12889-020-09810-2. PMID 33228625